CLINICAL TRIAL: NCT04064736
Title: Menstrual Health Interventions and School Attendance Among Ugandans
Acronym: MENISCUs-2
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ministry of Health, Uganda (Other Government); MRC/UVRI and LSHTM Uganda Research Unit (Other); WoMena Uganda (Unknown); Makerere University (Other); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: MENISCUs-2
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-08

CONDITIONS: Menstrual Health Intervention
Keywords: Menstrual Health; School attendance; Adolescent health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Management of menstruation can present substantial challenges to girls in low-income settings. The aim of this study is to pilot an intervention package to improve menstrual health (MH) management among school girls in 2 secondary schools in Entebbe sub-District, Uganda, and to prepare for a future cluster randomised trial to evaluate the impact of the intervention on school attendance, school performance and bacterial vaginosis.

The recently completed study (MENstrual hygiene and Safe male Circumcision in Ugandan Schools (MENISCUS-1) showed that menstruation is a key reason for school absenteeism in this setting. The qualitative research showed substantial embarrassment and fear of teasing regarding menstruation, and suggested that this, together with pain and lack of effective materials for menstrual hygiene management, led to school absenteeism. In a small quantitative sub-study of daily diaries, 40 girls reported school absence on 28% of period-days, compared with 7% of non-period days (adjusted odds ratio=5.99, 95%CI 4.4-8.2, p<0.001). Evaluation of menstrual management interventions, which address both the psycho social aspects of menstruation (knowledge, self-confidence, attitudes), and the physical aspects (management of pain, use of appropriate materials to eliminate leakage of menstrual blood, improved WASH facilities) are needed.

In the current study (MENISCUs-2), the investigators will pilot the MH interventions developed in MENISCUS-1 as a package delivered to all girls in one school year in two schools in Wakiso District. The intervention consists of:

* Training teachers to improve current delivery of the Government guidelines for puberty education delivered by teachers (usually female).
* A drama skit to address issues around menstruation, engaging girls, boys, parents and teachers.
* Provision of a menstrual management kit, including re-usable pads and training teachers and peers to teach girls how to use these menstrual management methods
* Supplying analgesics (paracetamol) for menstrual cramps using a voucher scheme
* Basic improvements to school sanitation facilities, including ensuring girls' privacy

The primary outcome is to review whether criteria for progression to a future trial are met. The criteria are that i) the education session and drama skit are delivered, the majority of girls use the pads, and that soap is available for >50% of observation visits; and ii) the retention rate in school over 9 months is >60%. The investigators will compare the relative risk of absenteeism on period-days and non-period-days from diaries, within MENISCUS-2 (the new pilot study in which the intervention will take place) and within MENISCUS-1 (the previous feasibility study where no intervention had taken place when the diaries were collected) schools. They will estimate the number of girls who are retained at school in order to estimate the likely loss to follow-up within a future trial. They plan to submit a proposal for a full trial in 2019.

DETAILED DESCRIPTION:
The study will take place in two secondary schools (one private and another government) in Entebbe sub-district. The study will take place among students in Class S2 aged. The study will consist of i) A stakeholder workshop to finalise the intervention including a Theory of Change workshop ii) Introduction of the intervention package to all S2 students and assess outcomes over 9 months (into the next school year), to assess retention (including those repeating year S2).

iii) Provision of daily diaries to a random sample of 50 students per school. A research assistant will make unannounced visits to the schools approximately every month to check the diaries and will collect them 2 weeks before the end of term (to avoid loss or damage).

iv) Cross-sectional surveys at baseline and endline in all girls in S2 to assess menstruation knowledge, attitudes, management practices and school absenteeism.

v) Cross-sectional surveys at baseline and endline for all boys in S2 to access menstruation attitudes and school absenteeism.

vi) Endline in-depth interviews (IDIs) will be conducted with 30 female students, 10 teachers (male and female) and 10 parents, sampled purposively (e.g. by attendance for girls) to assess perceptions of the interventions and impact on self-reported school absence vii) End line focus group discussions (FGDs) with two groups of girls in each school to assess their perceptions of the intervention and its impact on school attendance as well as one group of boys in each school to assess their perceptions of the intervention.

viii) Analysis of vouchers assessing uptake of analgesics ix) School examination data to assess performance x) Strengths & Difficulties questionnaire to assess psychosocial issues xi) Second stakeholder workshop will be held to discuss findings and plan for the future trial. This will include representatives from schools that are potential sites for the future trial.

Outcomes of the study: Primary outcome is school attendance using menstrual daily diaries for menstruating girls. School attendance will be compared using diaries, class registers, direct observation check visits and retrospective self-reported school attendance at the endline cross-sectional survey.

Secondary trial outcomes for the girls will be: 1) Knowledge and attitudes towards menstruation and MH evaluated using baseline and endline questionnaires with closed questions. Information will include menstruation knowledge and attitudes in boys and girls, and practices in girls; 2) Acceptability of re-usable pads (AFRIpads): In this trial development study, the study will provide girls with re-usable pads and collect further qualitative and quantitative data on the MH management methods practiced. To include girls' attitudes towards using the re-usable pads including privacy for changing and washing the re-usable pad. Ability to do usual activities and comfort or discomfort of use, ease of washing, drying and storing the re-usable pads, accessibility of water and soap, use of other MH methods alongside the re-usable pad, and feedback on the training given by WoMena the implementing partner.

3) Psychosocial issues: In the main trial the investigators will assess whether the intervention affects psychosocial outcomes through multiple methods including the quantitative interviews, the 25-item Strengths and Difficulties Questionnaire (self-report version; (http://www.sdqinfo.com) for 11-17 year-olds, and through qualitative methods. The SDQ consists of 25, 3-point Likert scale items from 0 'not true' to 2 'true', with a midpoint of 1 'somewhat true'.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were all male and female secondary students in the second school year in the 2 selecteed schools. Written informed consent was sought from students aged >18 years, and from the parents/caretakers of those aged <18 years, with student assent

Exclusion Criteria:

* None

Ages: 12 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: This pilot study was conducted in Entebbe Municipality in Wakiso District, Uganda. Entebbe has 13 registered secondary schools. Two day schools (one government and one private), both with students of low socio-economic status, were purposively selected.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
School attendance | 9 months
  Measured using menstrual daily diaries for menstruating girls. This will be compared using diaries, class registers, direct observation check visits and retrospective self-reported school attendance at the endline cross-sectional survey.

SECONDARY OUTCOMES:
Knowledge and attitudes towards menstruation | 9months
  Measured using baseline and endline questionnaires. Information included menstruation knowledge and attitudes in boys and girls, and practices in girls; 2) Acceptability of re-usable pads: In this trial development study, the investigators will provide girls with re-usable pads and collect further qualitative and quantitative data on the MH management methods practiced. To include girls' attitudes towards using the re-usable pads including privacy for changing and washing the re-usable pad. Ability to do usual activities and comfort or discomfort of use, ease of washing, drying and storing the re-usable pads, accessibility of water and soap, use of other MH methods alongside the re-usable pad, and feedback on the training on menstrual management given by WoMena the implementing partner.
Psychosocial wellbeing | 9months
  In the main trial the investigators propose to assess whether the intervention affects psychosocial outcomes through multiple methods including the quantitative interviews, the 25-item Strengths and Difficulties Questionnaire (self-report version; (http://www.sdqinfo.com) for 11-17 year-olds, and through qualitative methods. The SDQ consists of 25, 3-point Likert scale items from 0 'not true' to 2 'true', with a midpoint of 1 'somewhat true'.

CONTACTS AND LOCATIONS:
Locations (1):
- MRC/UVRI and LSHTM Uganda Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
: Data will be made available in the LSHTM Data Compass repository on request from the corresponding author (Helen Weiss https://orcid.org/0000-0003-3547-7936) from the website https://datacompass.lshtm.ac.uk/
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: From January 2020 with unlimited duration
URL: https://datacompass.lshtm.ac.uk/

REFERENCES:
- [Derived] Nalugya R, Tanton C, Hytti L, Kansiime C, Nakuya K, Namirembe P, Nakalema S, Neema S, Alezuyo C, Namuli Musoke S, Torondel B, Francis SC, Ross DA, Bonell C, Seeley J, Weiss HA. Assessing the effectiveness of a comprehensive menstrual health intervention program in Ugandan schools (MENISCUS): process evaluation of a pilot intervention study. Pilot Feasibility Stud. 2020 Apr 24;6:51. doi: 10.1186/s40814-020-00585-2. eCollection 2020. PMID 32346485
- [Derived] Kansiime C, Hytti L, Nalugya R, Nakuya K, Namirembe P, Nakalema S, Neema S, Tanton C, Alezuyo C, Namuli Musoke S, Torondel B, Francis SC, Ross DA, Bonell C, Seeley J, Weiss HA. Menstrual health intervention and school attendance in Uganda (MENISCUS-2): a pilot intervention study. BMJ Open. 2020 Feb 4;10(2):e031182. doi: 10.1136/bmjopen-2019-031182. PMID 32024786